CLINICAL TRIAL: NCT03012685
Title: Relationship Between Sleep the First Night and Week After Trauma and Subsequent Intrusive Memories: a Prospective Study From the Emergency Department
Brief Title: Sleep and Wellbeing Study
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Karolinska Institutet (Other); Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/EM/0326; 195832 (Other: IRAS)
Record Dates: First submitted 2016-10-25; First posted 2017-01-06 (Estimated); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sleep; Intrusive Memories; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Most people will experience a psychologically traumatic event, such as a life-threatening accident, at some point in their life. In the initial days after such an event, it is common to be haunted by intrusive memories: image-based memories of the event that spring to mind unbidden. Intrusive memories can be distressing in their own right, but are also a hallmark symptom of post-traumatic stress disorder (PTSD).

Sleep is important for many functions involved in how people perceive, respond to and remember events, including stressful/traumatic events. Studies with patients who have experienced traumatic events indicate that sleep disturbances in the first weeks post-trauma are associated with later PTSD symptoms. However, in a previous study with healthy volunteers exposed to experimental trauma (film footage), those who were sleep-deprived in the first night, compared to those who slept, had fewer intrusive memories in the following week. This raises the question of how sleep in the first night, but also the first week, after real-life trauma is related to subsequent intrusive memories and PTSD symptoms.

The current study is an observational study of patients recruited from a hospital emergency department after a traumatic event. After completing brief baseline questionnaires in the emergency department, participants will be asked to fill in a daily diary of their sleep and intrusive memories over the following week. Post-traumatic stress symptoms, anxiety and depression will be assessed by post/online at one week and two months. Participants will be telephoned after two months to complete an interview to assess PTSD symptoms and an optional feedback interview.

This clinical study will be the first to assess the relationship between sleep in the first night and week, and intrusive memories and mental wellbeing after real-life trauma. Findings may have implications for developing simple sleep-based preventive treatments after trauma in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Experienced or witnessed a traumatic event (i.e. one in which they were exposed to death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence)
* Present to the emergency department on the same day as the traumatic event
* Report memory of the event
* Fluent in written and spoken English
* Alert and orientated, Glasgow Coma Scale score (GCS) = 15
* Willing and able to give informed consent and complete study procedures

Exclusion Criteria:

* Loss of consciousness
* Current intoxication
* History of severe mental illness
* Current substance abuse or neurological condition
* Currently suicidal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the John Radcliffe Hospital Emergency Department after a traumatic event.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Daily diary of sleep and intrusive memories | 1 week

SECONDARY OUTCOMES:
Actigraphy - to assess sleep timing and duration | 1 week
Impact of Event Scale-Revised (total score and subscales scores) - to assess post-trauma distress | At 1 week and 2 months
Hospital Anxiety and Depression Scale | At 1 week and 2 months
Clinician-Administered PTSD Scale | At 2 months

OTHER OUTCOMES:
Feedback questionnaire | At 2 months
Optional feedback interview | After 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
It is planned to make an anonymised database available via the Open Science Framework

REFERENCES:
- [Background] Porcheret K, Iyadurai L, Bonsall MB, Goodwin GM, Beer SA, Darwent M, Holmes EA. Sleep and intrusive memories immediately after a traumatic event in emergency department patients. Sleep. 2020 Aug 12;43(8):zsaa033. doi: 10.1093/sleep/zsaa033. PMID 32133531